CLINICAL TRIAL: NCT05592379
Title: Consciousness and Psilocybin Effects on Well-Being (The CoPE Study): Pilot Phase
Brief Title: Consciousness, Psilocybin, and Well-Being
Acronym: CoPE Pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Usona Institute (Other); Tiny Blue Dot Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 2022-0746; A532017 (Other: UW Madison); Protocol Version 10/2/2024 (Other: UW Madison); 233897 (Other: OnCore ID)
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Psychedelic Experiences; Sleep
Keywords: Sleep; Psilocybin; Psychedelics; Healthy Volunteer
MeSH Terms: interventions — Psilocybin; Clonidine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: placebo first followed by placebo+clonidine or psilocybin+clonidine in asleep healthy volunteers
Who Masked: Participant
Masking Description: Participants may receive placebo (saline) or psilocybin during their treatment on overnight 2 but will not be told which they will receive.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1A: 2-minute IV Psilocybin+Clonidine / Saline in Asleep Participants (Experimental): Participants will receive 10 mL of placebo (saline) over 2 minutes while asleep during their first overnight visit. Participants will receive 0.2 mg oral clonidine and either 2 mg of IV psilocybin or saline over 2 minutes while asleep during their second overnight visit.
  Interventions: Drug: Psilocybin; Drug: Clonidine; Other: Saline
- Group 1B: 2-minute IV Psilocybin+Clonidine Infusion in Awake Participants (Experimental): If Group 1A participants can sleep 1 hour post-dosing and/or have no memory of dosing, Group 1B moves forward and participants will receive 0.2 mg clonidine and 2 mg of IV psilocybin over 2 minutes while awake.
  Interventions: Drug: Psilocybin; Drug: Clonidine
- Group 2A: 2-minute IV Psilocybin+Clonidine / Saline in Asleep Participants (Experimental): If Group 1A participants fail to sleep 1 hour post-dose, Group 2A moves forward. Participants will receive 10 mL of placebo (saline) over 10 minutes while asleep during their first overnight visit. Participants will receive 0.2 mg oral clonidine and either 2 mg of IV psilocybin or saline over 10 minutes while asleep during their second overnight visit.
  Interventions: Drug: Psilocybin; Drug: Clonidine; Other: Saline
- Group 2B: 10-minute IV Psilocybin+Clonidine in Awake Participants (Experimental): If Group 2A participants can sleep 1 hour post-dosing and/or have no memory of dosing, Group 2B moves forward and participants will receive 0.2 mg clonidine and 2 mg of IV psilocybin over 10 minutes while awake.
  Interventions: Drug: Psilocybin; Drug: Clonidine
- Group 1C: 2-minute IV Psilocybin Alone in Awake Participants (Active Comparator): If Group 1A allows for sleep 1 hour post dose, Group 1C will move forward and participants will receive 2mg of IV psilocybin over 2 minutes while awake for comparison.
  Interventions: Drug: Psilocybin
- Group 2C: 10-minute IV Psilocybin Alone in Awake Participants (Active Comparator): If Group 2A allows for sleep 1 hour post dose, Group 2C will move forward and participants will receive 2mg of IV psilocybin over 10 minutes while awake for comparison.
  Interventions: Drug: Psilocybin
- Initial Groups 1A and 2A (Experimental): Participants will receive 2mg of IV psilocybin over 2 minutes or 10 minutes while asleep during an overnight visit and 10 mL of placebo (saline) over 2 minutes or 10 minutes while asleep during another overnight visit. The order of administration will be determined by the study protocol.
  Interventions: Drug: Psilocybin; Other: Saline

INTERVENTIONS:
Drug: Psilocybin — The IV formulation of psilocybin will be prepared using bulk psilocybin that will satisfy Good Manufacturing Practice (GMP) criteria. The IV psilocybin solution will be prepared under sterile conditions by the University of Wisconsin Pharmaceutical Research Center (PRC).
  Other Names: Psilocybine; Psilocibin
Drug: Clonidine — Clonidine will be administered orally in a 0.2mg dose
  Arms: Group 1A: 2-minute IV Psilocybin+Clonidine / Saline in Asleep Participants; Group 1B: 2-minute IV Psilocybin+Clonidine Infusion in Awake Participants; Group 2A: 2-minute IV Psilocybin+Clonidine / Saline in Asleep Participants; Group 2B: 10-minute IV Psilocybin+Clonidine in Awake Participants
Other: Saline — The IV placebo (saline) will be prepared under sterile conditions by the University of Wisconsin Pharmaceutical Research Center.
  Other Names: Placebo
  Arms: Group 1A: 2-minute IV Psilocybin+Clonidine / Saline in Asleep Participants; Group 2A: 2-minute IV Psilocybin+Clonidine / Saline in Asleep Participants; Initial Groups 1A and 2A

SUMMARY:
This study is being done to identify a dosing strategy that will allow IV psilocybin to be administered to sleeping participants without awakening them.

DETAILED DESCRIPTION:
The study commenced with 1 subject receiving 2 mg IV infusion of psilocybin over 2 minutes and 2 subjects receiving 2 mg IV infusion of psilocybin over 10 minutes. Subsequently, the pre-treatment of 0.2 mg of clonidine was added.

This design involves testing up to two psilocybin+clonidine administration protocols in asleep and awake subjects and one of two "IV psilocybin only" administration protocols in awake subjects.

The updated protocol entails 2 mg of psilocybin administered via IV infusion combined with 0.2 mg oral clonidine in sleeping subjects. If either the 2-minute or 10-minute psilocybin infusion (plus oral clonidine) protocols allow sleep maintenance, up to 5 subjects will, while awake, receive the same psilocybin infusion protocol administered to sleeping subjects, including clonidine. Subsequently, this same infusion protocol may be administered without clonidine, to evaluate any potential effect of co-administered clonidine on the acute psychedelic experience in awake subjects (Group 1C for 2-minute psilocybin infusion; Group 2C for 10-minute psilocybin infusion), should a significant effect of clonidine on the awake psychedelic experience be suspected. For individual subjects that are dosed first while asleep and then up to twice while awake, each of their visits will be separated by a minimum of two weeks and will include psychosocial support through integration sessions following each dosing visit.

Adaptive Study Design Change per Protocol Amendment Approved 5/21/24

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy
* English-speaking
* Live within 150 miles of Madison, WI for duration of study

Exclusion Criteria:

* Current use of medications that may interact with psilocybin
* Current sleep disorder, including (but not limited to) insomnia, sleep apnea, restless legs syndrome, and/or narcolepsy
* Females with positive urine pregnancy at any time point during screening or study participation
* Current cardiac valve disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Number and nature of adverse events associated with the administration of a single dose of IV psilocybin | Up to 9 days
  Adverse events associated with the administration of a single dose of IV psilocybin administered either alone or in combination with oral clonidine in asleep and awake participants. Adverse event grading will be done using Common Terminology Criteria for Adverse Event (CTCAE)Adverse events will be graded from Grade 1-5 depending on severity. Grade 1 - mild, grade 2 - moderate, grade 3 - severe, grade 4 - Life threatening, grade 5 - Fatal. Adverse events will be collected on an Adverse Event Log throughout the study.

SECONDARY OUTCOMES:
Number of participants administered psilocybin plus clonidine while asleep who remain asleep for at least 1 hour post dosing and/or report no memory of the dosing experience upon awakening | 1 day
Post-dosing scores on the 30-item Mystical Experiences Questionnaire (MEQ30) following administration of psilocybin and clonidine while asleep or awake | 1 day
  The MEQ30 is a 30-item self-report measure developed to assess the effects of classic psychedelics in laboratory studies. It covers the major dimensions of the classic mystical experience: unity, transcendence, noetic quality, sacredness, positive mood, and ineffability/paradoxicality. The MEQ has 4 sub scales: 1) transcendence, 2) positive mood, 3) ineffability, and 4) mystical. The total possible range for each sub scale and total score is 0-100% with higher percentages indicating a larger mystical experience. Typically, a complete mystical experience is defined as scoring 60% or more on all four MEQ30 subscales.
Post-dosing scores on the Emotional Breakthrough Inventory (EBI) following administration of IV psilocybin either alone or in combination with clonidine while awake | 1 day
  The EBI is a 6-item self-report scale that assesses the presence and severity of emotionally challenging/distressing experiences that occur during a psychedelic experience. The scale utilizes visual analog responses captured on a line anchored by "not at all" on one end and "very much so" on the other. Experiences queried include 1) facing emotionally difficult feelings that are usually pushed aside; 2) experiencing a resolution of a personal conflict/trauma; 3) being able to explore challenging emotions and memories; 4) having an emotional breakthrough; 5) getting a sense of closure on an emotional problem, and 6) achieving an emotional release followed by a sense of relief. The total possible range of scores for the EBI is 0-100 with higher scores indicating a greater emotional breakthrough.
Post-dosing scores on the Psychological Insight Scale (PIS) following administration of IV psilocybin either alone or in combination with clonidine while awake | 1 day
  The PIS is a 6-item self-report scale that queries the acquisition of insight following a psychedelic therapy. The items are answered with visual analogue scales anchored by "no more than usually" on the left and "much more than usually" on the far right. A seventh item separately assesses self-reported behavioral change resulting from the psychedelic experience. The total possible range of scores for the PIS is 0-100 with higher scores indicating a greater psychological insight.
Post-dosing scores on the Ego Dissolution Inventory (EDI) following administration of IV psilocybin either alone or in combination with clonidine while awake | 1 day
  The EDI is an 8-item self-report scale designed to measure ego-dissolution. Each item is scored on a visual analogue scale from 0 to 100 with the following statements at the lower and upper end, respectively: "No, not more than usually" and "Yes, I experienced this completely/entirely." The total possible range of scores for the EDI is 0-100 with higher scores indicating a greater ego dissolution.
Post-dosing scores on the Awe Experiences Scale (AWE) following administration of IV psilocybin either alone or in combination with clonidine while awake | 1 day
  The AWE is a 30-item self-report scale that measures the state of awe. Each items is rated on a scale of 1 to 7, with 1 representing "Strongly Disagree" and 7 representing "Strongly Agree". The total possible range of scores for the AWE is 1-7 with higher scores indicating a greater awe.
Post-dosing scores on the Altered States of Consciousness Questionnaire (ASC) following administration of IV psilocybin while either alone or in combination with clonidine while awake | 1 day
  The ASC is a 94-item self-report scale that assesses alterations from your normal waking consciousness. Each item is scored on a visual analogue scale from 0 to 100 with the following statements at the lower and upper end, respectively: "No, not more than usually" and "Yes, much more than usually." The total possible range of scores for the ASC is 0-100 with higher scores indicating a greater state of altered consciousness.
Post-dosing scores on the Challenging Experiences Questionnaire (CEQ) following administration of IV psilocybin either alone or in combination with clonidine while awake | 1 day
  The CEQ is a 26-item questionnaire that consists of seven factors of challenging experience with psilocybin mushrooms: fear, grief, feeling of losing your sanity (insanity), feel as though you are dying (death), feelings of isolation, physiological distress, and paranoia. The CEQ uses a 6-point response scale [0: None/not at all, 1: So slight cannot decide, 2: Slight, 3: Moderate, 4: Strong; 5: Extreme (more than ever before in my life)] to indicate the degree to which a participant experiences each of a series of subjective effects during their psilocybin session. Total CEQ score is expressed as the percentage of the total possible ratings on the scale. The total possible range of scores for the CEQ is 0-5 with higher scores indicating a greater challenging experience.
Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) score 7 days post administration of IV psilocybin either alone or in combination with clonidine while awake | Up to 19 days
  The WEMWBS is a 14-item self-report scale that was designed to measure the psychological well-being of a population. The questions use a five-point Likert scale. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing. Items on the questionnaire are rated on a 5-point scale, where 1= "None of the time", 2= "rarely", 3= "some of the time", 4= "often", 5= "all the time". A total scale score is calculated by summing the 14 individual item scores. The total possible range of scores for the WEMWBS is 14-70 with higher scores indicating a greater well-being.
World Health Organization Well-Being Index | Up to 19 days
  World Health Organization Well-Being Index (WHO-5) is a 5-item survey with a total possible range of scores 0-25 where higher scores indicate increased well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
IDP will not be made available to other researchers.